CLINICAL TRIAL: NCT01410994
Title: Study of Renal Parameters After Bariatric Surgical Weight Loss
Brief Title: Bariatric Surgery and the Kidney
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Allon Friedman, MD, Assistant Professor, Indiana University
Other Study IDs: 1102-06
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Proteinuria
Keywords: glomerular filtration rate
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the project is to study the relationship between post-bariatric surgery changes in weight and renal parameters.

ELIGIBILITY:
Inclusion Criteria:

* bariatric patients

Exclusion Criteria:

* age <18
* dialysis dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: bariatric surgery patients in the Indianapolis region
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
GFR | April 2014

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Indianapolis, Indiana, United States